CLINICAL TRIAL: NCT06407869
Title: Effects of Functional Progressive Strength Training on Gait Parameters and Walking Capacity in Children With Spastic Cerebral Palsy
Brief Title: Effects of Functional Progressive Strength Training in Children With Spastic Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: REC/RCR&AHS/23/0778
Record Dates: First submitted 2024-05-06; First posted 2024-05-09 (Actual); Last update posted 2024-10-28 (Actual); Status verified 2024-10

CONDITIONS: Spastic Cerebral Palsy
Keywords: Spastic CP, Functional Progressive Strength Training
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Intervention Model Description: It will be randomized control trial in which random sampling technique will be used. Two groups of 6-12 age will be formed in which participants will randomly be divided. Group A will receive Functional Progressive Resistance Exercises and group B will receive conventional stretching and strengthening exercises
Who Masked: Participant
Masking Description: Participants will get separate treatment protocols and possible efforts will be put to mask both groups about treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Functional Progressive Strength Training (Experimental): group of 20 children with spastic cerebral palsy on which FPST techniques including 3 or 4 PRT sessions per week for 12 weekswill be applied.
  Interventions: Other: Functional Progressive Strength Training
- Control (Other): group of 20 children with spastic cerebral palsy on which conventional physical therapy techniques will be applied
  Interventions: Other: Control

INTERVENTIONS:
Other: Functional Progressive Strength Training — The Functional Progressive Resistance Exercise (FPRE) protocol is designed to improve functional strength through structured workouts. It begins with a 3-minute warmup involving stretching and range of motion exercises, followed by progressively intense sit-to-stand exercises over six weeks. Participants also perform half-kneeling, standing up, and side-step-up exercises, with 20 minutes of total activity and rest intervals. The session ends with a 2-minute cooldown. Weights are gradually increased up to 15 times the initial load, with a minimum of one-minute rest between sets. The regimen is tailored through trial and error to find the maximum load participants can effectively manage.
  Arms: Functional Progressive Strength Training
Other: Control — conventional physical therapy techniques will be applied
  Arms: Control

SUMMARY:
This study focuses on the effects of Functional Progressive Strength Training (FPST) on children with spastic cerebral palsy, a condition characterized by increased muscle tone that affects movement. Spastic cerebral palsy is one type of cerebral palsy, with others including dyskinetic, which involves involuntary movements, and ataxic, which affects coordination. FPST differs from traditional strength training by incorporating exercises that replicate everyday activities to integrate strength use in daily movements. The study uses an experimental design with participants aged 6-12 years, recruited from specialized centers. They are randomly assigned to either a treatment group receiving FPST or a control group receiving standard care. The study aims to measure improvements in gait and mobility, assessed through various tools like step and stride length, cadence, and gait speed, alongside caregiver reports and direct observations. Statistical analyses will determine the effectiveness of FPST in enhancing motor function and walking capacity in these children.

DETAILED DESCRIPTION:
In the outlined study, participants who fit the necessary inclusion and exclusion criteria are asked to provide written informed consent before taking part. The randomization process involves each participant drawing a number from a box: those who draw number one are placed in Group A (experimental group), while those drawing number two are placed in Group B (control group).

Group A undergoes a specialized treatment approach called Functional Progressive Resistance Exercise (FPRE), in addition to receiving conventional treatment. The FPRE regimen starts with a three-minute warm-up that includes range of motion mobilization and stretching exercises. This is followed by a series of resistance exercises, such as sit-to-stand activities, which increase in intensity over a six-week period, targeting specific percentages of body weight. The participants then engage in half-kneeling, standing up, and side-step-up exercises for 20 minutes each, with rest intervals. The session concludes with a two-minute cooldown. The protocol is designed to gradually increase the load carried by the participants, scaling up to five times, then 10 times, and eventually 15 times the initial weight, with a minimum of one minute of rest between sets. The exercises are calibrated through trial and error to find the maximum load that can be lifted for the defined number of repetitions and sets.

Group B participants receive conventional physical therapy aimed at maintaining muscle flexibility and improving motor function. Their routine includes an hour-long session three times a week, consisting of stretching exercises focused on muscles prone to tightness, such as the Achilles tendons, hamstrings, hip flexors, and adductors. Strength training targets specific muscle groups including hip flexors, knee extensors, and ankle dorsiflexors. The gait training in Group B starts in a controlled environment, such as walking between parallel bars, and progresses to more complex tasks like walking unassisted in open spaces, navigating different floor surfaces, and moving through obstacle-laden paths.

Both groups are reassessed after 12 weeks to evaluate the impact of their respective interventions on gait parameters and walking capacity, using a combination of direct observation, caregiver reports, and standardized assessment tools. The study aims to ascertain the relative efficacy of these two approaches in enhancing mobility and quality of life for children with spastic cerebral palsy.

ELIGIBILITY:
Inclusion Criteria:

* Aged 6 to 12 years
* Children had to be able to understand and follow instructions
* Diplegic CP
* GMFSC I, II, III

Exclusion Criteria:

* Treatment with botulinum toxin A in lower limb.
* Rhizotomy done 6 months before the study.
* Children with unstable seizures will be excluded.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2024-06-28 (Actual); Primary Completion 2024-08-20 (Actual); Study Completion 2024-08-25 (Actual)

PRIMARY OUTCOMES:
Gait Parameters | 12 weeks
  To assess gait parameters in a study, four tools are utilized: step length, measuring the distance between alternating heel strikes; stride length, measuring the distance between two heel strikes of the same extremity; cadence, counting the number of steps taken; and gait speed, timing the duration to cover a 5-meter distance with a stopwatch.

SECONDARY OUTCOMES:
1-Minute Walk Test | 12 weeks
  The 1-minute walk test assesses walking capacity on a 20-meter indoor track, recording the distance a participant covers in one minute while walking as fast as possible without running.

CONTACTS AND LOCATIONS:
Overall Officials: Kashaf Naeem, MS*, Principal Investigator — Riphah International University
Locations (1):
- Riphah International University, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hanssen B, Peeters N, De Beukelaer N, Vannerom A, Peeters L, Molenaers G, Van Campenhout A, Deschepper E, Van den Broeck C, Desloovere K. Progressive resistance training for children with cerebral palsy: A randomized controlled trial evaluating the effects on muscle strength and morphology. Front Physiol. 2022 Oct 4;13:911162. doi: 10.3389/fphys.2022.911162. eCollection 2022. PMID 36267577